CLINICAL TRIAL: NCT03342495
Title: Evaluating Innovations in Transition From Pediatric to Adult Care - The Transition Navigator Trial
Acronym: TNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB16-2561
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Endocrine System Diseases; Gastro-Intestinal Disorder; Neuro-Degenerative Disease; Epilepsy; Autoimmune Diseases; Renal Disease; Cardiac Disease; Metabolic Disease; Genetic Diseases, Inborn; Respiratory Disease; Hematologic Diseases; Autism Spectrum Disorder; Fetal Alcohol Spectrum Disorders; Traumatic Brain Injury; Stroke
Keywords: transition, young adults, transfer
MeSH Terms: conditions — Diabetes Mellitus; Endocrine System Diseases; Digestive System Diseases; Epilepsy; Autoimmune Diseases; Kidney Diseases; Heart Diseases; Metabolic Diseases; Genetic Diseases, Inborn; Respiration Disorders; Hematologic Diseases; Autism Spectrum Disorder; Fetal Alcohol Spectrum Disorders; Brain Injuries, Traumatic; Stroke | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Two groups of participants will be randomized by primary clinical area
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigator Arm (Experimental): Patient Navigator (Social Worker) will assist youth adapt and attach to adult delivered healthcare for up to 24 months.
  Participants will receive 5 issues of a provincial generic newsletter on topics around transition.
  Participants will be asked to complete a health questionnaire at baseline and 4 more times during 24 months.
  Participants will be asked to complete a transition readiness questionnaire at baseline and 4 more times during 24 months.
  Participants will be provided the opportunity to journal online about their experiences.
  Up to 100 participants will be provided the opportunity to be interviewed at baseline and end of study about their transition experience.
  Interventions: Other: Patient Navigator
- Usual Care Arm (Other): Youth will receive usual care from their pediatric clinics in preparation and transfer to adult care.
  Participants will receive 5 issues of a provincial generic newsletter on topics around transition.
  Participants will be asked to complete a health questionnaire at baseline and 4 more times during 24 months.
  Participants will be asked to complete a transition readiness questionnaire at baseline and 4 more times during 24 months.
  Participants will be provided the opportunity to journal online about their experiences.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Patient Navigator — Social worker/Patient Navigator will be assigned to follow youth in adult care for up to 24 months to assist youth adapt and attach to adult delivered healthcare
  Arms: Patient Navigator Arm
Other: Usual Care — Whatever processes are in place in a variety of clinics to support transfer from pediatric to adult care in the pediatric clinics
  Arms: Usual Care Arm

SUMMARY:
The Transition Navigator Trial (TNT) is a pragmatic randomized controlled trial evaluating the effectiveness of usual care plus a patient navigator service versus usual care plus newsletters and other educational materials, to improve transition outcomes among adolescents aged 16-21 who have chronic health conditions requiring transfer to adult specialty care.

The study will provide urgently needed data to guide health care providers and policy makers regarding the provision of coordinated transition care. These results have the potential to:

1. Change care delivery
2. Improve health outcomes
3. Improve the experiences of young adult transition to adult care

DETAILED DESCRIPTION:
Transition is the purposeful, planned movement of adolescent and young adults with chronic health conditions from child-centered to adult-oriented health systems. Transition includes, but is not limited to transfer to adult care. Transfer of care, which occurs during a vulnerable developmental period around age 18 introduces gaps in continuity of care that can lead to detrimental health outcomes in young adults. Therefore, provision of coordinated and developmentally appropriate care during the transition period is necessary to maintain health and to sustain investments made in pediatric health care.

Clinical practice guidelines for transition to adult care recommend the use of patient navigators to coordinate the entry of patients into a complex and unfamiliar adult health care system. Patient navigators provide individualized supports to facilitate medical follow-up and adherence. A limited number of studies have shown that access to a patient navigator during transition decreases drop-out from medical care and disease specific adverse events. No study to date has evaluated the benefits of a patient navigator to improve patient and or health system outcomes, when implemented across multiple chronic disease settings.

Objectives/Methods

1. to evaluate the impact of a patient navigator intervention compared to treatment as usual for 16 to 21 year olds living with chronic health conditions who are transferring to adult care with respect to healthcare utilization and patient reported outcomes
2. to obtain perceptions of stakeholders regarding the role of patient navigators in reducing barriers to adult-oriented ambulatory care
3. to determine the net health care cost impact attributable to the navigator intervention

A qualitative study sampling participants randomized into the intervention arm at the beginning and end of the trial will also be undertaken to understand the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* has a chronic medical condition (defined as conditions which are >3 months in duration and/or lifelong with multiple morbidities and/or multi-organ/system manifestations or condition with typically affect a single organ/system), who are expected to be transferred to adult specialty follow-up
* Last planned pediatric visit within up to 12 months after assessment of eligibility

Exclusion Criteria:

* cannot consent in English
* moving out of province within 24 months
* enrolled in another transition navigator study

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 337 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Health services utilization | 12 to 24 months
  verification of health services utilized by up to 600 participants collected via personal health numbers (e.g. National Ambulatory Care Reporting System; Alberta Ambulatory Care Reporting System; Discharge Abstract Database; Physician Claims)

SECONDARY OUTCOMES:
cost analysis | up to 24 months
  did the intervention save high cost service provision
Variation in TRAQ (Transition Readiness Questionnaire) scores | Enrollment and 3 subsequent times in 24 months
  Variation in TRAQ scores; comparing intervention and non-intervention arm
Variation in SF-12 Scores | Enrollment and 3 subsequent times in 24 months
  Participant reported mental and physical health

OTHER OUTCOMES:
Youth/Caregiver Satisfaction | after 12 to 24 months
  Qualitative Interviews with sampling of participants from patient navigator intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Susan Samuel, MD, MSc, Principal Investigator — University of Calgary; Gina Dimitropoulos, PhD, Principal Investigator — University of Calgary; Andrew Mackie, MD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Stollery Childrens Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samuel S, Punjwani Z, San Martin-Feeney D, Allemang B, Guilcher GMT, Lang E, Pacaud D, Pinzon J, Andrew G, Zwaigenbaum L, Perrott C, Andersen J, Hamiwka L, Nettel-Aguirre A, Klarenbach S, McBrien K, Scott SD, Patton M, Samborn S, Pfister K, Ryan L, Dimitropoulos G, Mackie AS. Effectiveness of Patient Navigation During Transition to Adult Care: A Randomized Clinical Trial. JAMA Pediatr. 2025 Apr 1;179(4):375-382. doi: 10.1001/jamapediatrics.2024.6192. PMID 39928304
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Samuel S, Dimitropoulos G, Schraeder K, Klarenbach S, Nettel-Aguirre A, Guilcher G, Pacaud D, Pinzon J, Lang E, Andrew G, Zwaigenbaum L, Scott S, McBrien K, Hamiwka L, Mackie A. Pragmatic trial evaluating the effectiveness of a patient navigator to decrease emergency room utilisation in transition age youth with chronic conditions: the Transition Navigator Trial protocol. BMJ Open. 2019 Dec 10;9(12):e034309. doi: 10.1136/bmjopen-2019-034309. PMID 31826899